CLINICAL TRIAL: NCT01690754
Title: Monitoring Patient Compliance With Tuberculosis Treatment Regimens
Brief Title: Evaluating the Effectiveness of Interactive SMS Reminders on TB Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interactive Research and Development (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Shama Mohammed, Associate Researcher, Interactive Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRD_IRB_2011_03_002
Record Dates: First submitted 2012-09-13; First posted 2012-09-24 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Tuberculosis
Keywords: SMS; tuberculosis; impact evaluation
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This arm will receive the regular standard of care given by TB clinics.
- Interactive Reminders (Experimental): Patients randomized to this arm will receive Interactive SMS reminders daily.
  Interventions: Other: Interactive Reminders

INTERVENTIONS:
Other: Interactive Reminders — Daily SMS reminders sent to TB patients at a pre-specified time. They are asked to respond to the reminders. If a response is not received within two hours, they are sent another reminder for up to three per day.
  Arms: Interactive Reminders

SUMMARY:
In this study, Interactive Research and Development (IRD) in Karachi, Pakistan is evaluating the impact of Interactive Reminders on drug compliance and treatment outcomes. Interactive Reminders is an interactive SMS reminder system to help patients remember to take their TB medication. In this system, patients receive daily SMS reminders for the duration of their treatment at a pre-specified time, reminding them to take their medication. Patients are asked to reply back to the system, either through SMS or a missed call, with the time they took their medicine that day. If a response is not received within two hours, a second reminder is sent. If a response is still not received in a further two hours, a third and final reminder for the day is sent. Non-responsive patients are followed up with phone calls and a list of non-responsive patients is shared with clinics based on the parameters of non-responsiveness that they specify.

IRD seeks to determine the impact of this system on treatment outcomes and compliance to prescribed medication through administering a randomized control trial among newly diagnosed TB patients in Karachi, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* New, smear-positive drug susceptible TB who have been on treatment for less than two weeks
* Access to a mobile phone (self-reported)
* Intending to reside in Karachi for the duration of their treatment

Exclusion Criteria:

* Patients who do not have regular access to a mobile phone
* Patients who have previously received TB treatment
* Patients who have another member in their household who is already a part of the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2207 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Treatment Outcomes | After 6 to 8 months of treatment
  The investigators will compare clinically reported treatment outcomes between the intervention and control groups.

SECONDARY OUTCOMES:
Physical fitness and mobility | Monthly visits for 6 to 8 months of treatment
  The investigators will measure physical fitness and mobility through questionnaires conducted with patients during household visits each month that they are on treatment. The investigators are using two indices. The physical fitness index will record respondents ability to perform certain tasks. The mobility index will record the mobility of participants.
Psychological Impacts | Monthly visits for 6 to 8 months of treatment
  In order to gauge the psychological impacts of the system, the investigators will be looking at participants' perceptions on the likelihood of being cured, how they feel on a given day using the pain scale, and how supported they feel. This data will be collected through questionnaires conducted at each monthly mid-line visit.
Self-reported medication adherence | "Surprise" monthly visits during treatment
  Medication adherence will be measured through self-reports by participants on whether they took their TB medication in the past 24 hours. This data will be collected through monthly "surprise" visits to the participants' houses.
Sputum conversion | At 1, 2, 5, and 6/7 months of treatment
  The investigators will look at sputum test results for patients at months 2, 5, and 6/7 of their treatment to compare when sputum conversion occurs between the intervention and control group at these three periods during their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Glennerster, PhD., Principal Investigator — Massachusetts Institute of Technology; Shama Mohammed, MPA/ID, Principal Investigator — Interactive Research and Development; Aamir J. Khan, MD/PhD., Principal Investigator — Interactive Research and Development
Locations (11):
- Pakistan (11):
  - Civil Hospital, Karachi
  - Indus Hospital, Karachi
  - Jinnah Postgraduate Medical Center, Karachi
  - Landhi Medical Complex, Karachi
  - Private GP clinics and Private labs partnering with Interactive Research and Devellopment, Karachi
  - Sindh Government Hospital - Liaqatabad, Karachi
  - Sindh Government Hospital - New Karachi, Karachi
  - Sindh Government Hospital - Qatar, Karachi
  - Sindh Government Hospital New Karachi Kaali Market, Karachi
  - UHC-New Karachi, Karachi
  - Urban Health Center - Landhi, Karachi

REFERENCES:
- [Derived] Mohammed S, Glennerster R, Khan AJ. Impact of a Daily SMS Medication Reminder System on Tuberculosis Treatment Outcomes: A Randomized Controlled Trial. PLoS One. 2016 Nov 1;11(11):e0162944. doi: 10.1371/journal.pone.0162944. eCollection 2016. PMID 27802283